CLINICAL TRIAL: NCT03848533
Title: Effect of the Administration of Melatonin and Metformin on Glycemic Control, Genotoxicity and Cytotoxicity Markers in Patients With Prediabetes: Pilot Study
Brief Title: Effect of Melatonin and Metformin on Glycemic Control Genotoxicity and Cytotoxicity Markers in Patients With Prediabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Lizet Yadira Rosales Rivera, Profesor investigador asociado C, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-MEL-LESM
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-02

CONDITIONS: PreDiabetes
Keywords: Melatonin; Metformin; Pre Diabetes; PreDiabetes; Micronuclei; Genotoxicity Markers; Cytotoxicity Markers
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Melatonin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: It will be done using a sealed envelope, which will contain a letter A, B or C, and will be given to choose an envelope to the participants. The letter obtained will indicate the group to which the subject will belong during the intervention. The intervention designated for each of the groups will be unknown by the researcher and participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- melatonin plus metformin (Experimental): It will be indicate metformin 850 mg tablets, once a day in the morning (before breakfast) per 90 days.
  Will administrate melatonin 5 mg lengthed release capsules, once a day in the night (before bedtime) per 90 days.
  Interventions: Drug: melatonin; Drug: metformin
- metformin plus placebo (Active Comparator): It will be indicate metformin 850 mg tablets, once a day in the morning (before breakfast) per 90 days.
  Will administrate homologated placebo once a day in the night (before bedtime) per 90 days.
  Interventions: Drug: metformin; Drug: Placebo
- melatonin plus placebo (Experimental): It will be indicate homologated placebo once a day in the morning (before breakfast) per 90 days.
  Will administrate melatonin 5 mg lengthed release capsules, once a day in the night (before sleep) per 90 days.
  Interventions: Drug: melatonin; Drug: Placebo

INTERVENTIONS:
Drug: melatonin — The administration of melatonin will be indicated at night before bedtime to avoid alterations of the circadian cycle. It will be contained in bottles labeled "Medication 2" to maintain the masking. This intervention will be indicated in two groups (Melatonin plus metformin and Melatonin plus placebo)
  Other Names: Cronocaps
  Arms: melatonin plus metformin; melatonin plus placebo
Drug: metformin — For the intervention with metformin, prolonged-release tablets will be used to reduce adverse effects and improve adherence to treatment. It will be contained in bottles labeled "Medication 1" to maintain masking. This intervention will be indicated in two groups (Melatonin plus metformin and metformin plus placebo)
  Other Names: Ifor
  Arms: melatonin plus metformin; metformin plus placebo
Drug: Placebo — The placebo may be contained in bottles labeled "Medication 1" or "Medication 2" depending on the time of administration, and the group in which it is used. Placebo will be used in two groups (Melatonin plus placebo and Metformin plus placebo)
  Other Names: Calcined magnesia
  Arms: melatonin plus placebo; metformin plus placebo

SUMMARY:
Melatonin is a hormone that regulates the circadian cycle in addition to having an antioxidant effect. Patients with prediabetes state, has a deregulation of glucose metabolism and an overproduction of reactive oxygen species caused by levels of hyperglycemia that generate DNA modification in pancreatic beta cells, which leads to apoptosis and a deficient production of insulin. The administration of metformin and melatonin could be a possibility to treat and reverse the prediabetic state decreasing the glycemic levels and reactive oxygen species production.

DETAILED DESCRIPTION:
A randomized, double blind, placebo-controlled, pilot clinical trial will carried out in 42 patients with a diagnosis of prediabetes, according to the American Diabetes Association criteria. The patients will be divide in three groups administrating metformin plus placebo, melatonin plus placebo or melatonin plus metformin. The intervention will be with 500 mg lengthed release tablets of metformin once a day in the morning, per 90 days, 5 mg lengthed release capsules of melatonin one a day in the night per 90 days and calcined magnesia as a placebo. Before and after the intervention, will be evaluate: fasting plasma glucose, blood glucose after an oral glucose tolerance test, A1c hemoglobin fraction, micronuclei frequency, nuclear anomalies frequency, insulin secretion and insulin sensitivity, weight, height, body mass index, triglycerides, total cholesterol, high-density lipoprotein, low-density lipoprotein, creatinine, uric acid, and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Age beween 30 to 60 years old.
* Diagnosis of Prediabetes state according to the American Diabetes Association criteria.
* Without pharmacological treatment.
* Body mass index between 25 to 34.9 Kg/m2
* Sign informed consent

Exclusion Criteria:

* Patients with pharmacological treatment.
* Pregnant woman
* Patients with autoimmune, cancer, reumatic diases history or with pharmaceutical treatment
* Workers on night or changing shifts.
* Subjects that have been exposed to radiation
* Dyslipidemia: Total cholesterol >250mg/dL, Triglycerides >500 mg/dL.
* Subjects that have travel to other place with a different time zone.
* Patients with diagnosis of insomnia
* Patients with a glomerular filtration <60 ml/min using the Cockroft-Gault Formula.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG) | Baseline to week 12
  The FPG will be evaluate in a blood sample after a 8 - 12 hour fasting period. Will be use a fotometric quantification of glucose levels in plasma sample and will report in mg/dL.
Blood Glucose level after an Oral Glucose tolerance Test | Baseline to week 12
  Will estimate the glucose levels at 2 hours after administration of 75 grams of anhydrid dextrosa. The result will report in mg/dL.
A1c Hemoglobin Fraction (HbA1C) | Baseline to week 12
  HbA1c will be measured with High-performance liquid chromatography technique from a blood sample. The result will report in percentage (%).
Micronuclei frequency | Baseline to week 12
  The frequency of micronuclei will be measured from a cytological sample obtained from the oral epithelium by careful scraping of both cheeks. A fluorescence technique will be performed using acridine orange, as well as a Giemsa-Wrigth stain. The result will be reported in micronucleus frequency per 1000 cells.
Nuclear anomalies frequency | Baseline to week 12
  The nuclear anomalies frequency will be measured from a cytological sample obtained from the oral epithelium by careful scraping of both cheeks. A fluorescence technique will be performed using acridine orange, as well as a Giemsa-Wrigth stain. They will be divided according to their morphology (multinucleated cells, pyknotic nucleus, karyorrhexis, caryolysis, nuclei buds, condensed chromatin) and will be reported by the number of findings per 1000 cells.

SECONDARY OUTCOMES:
Body height | Baseline to week 12
  It will be determined using the electric bioimpedance scale with electrical stadiometer. The measurement will be made with the patient standing on the marks on the bioimpedance scale, in an upright position. This determination will be reported in meters (m) with a minimum precision of 0.01 meters.
Body weight | Baseline to week 12
  t will be determined using the electric bioimpedance scale with electrical stadiometer. The measurement will be made with the patient standing on the marks on the bioimpedance scale, in an upright position. This determination will be reported in kilograms (Kg).
Body mass index | Baseline to week 12
  The calculation will be made using the results of the weight, and height. From these results will be calculated by dividing the weight obtained over the square of the height. This index will be reported in kilograms per square meter (kg / m2)
Insulin Secretion | Baseline to week 12
  The calculation will be made using the insulogenic index, using the values obtained in the oral glucose tolerance test, and determining the insulin levels in plasma at 120 minutes and at the baseline measurement, as well as the glucose levels obtained at the 120 minutes and at the baseline measurement.
Baseline Insulin Secretion | Baseline to week 12
  It will be use the Stumvoll index for the calculation of this parameter.
Insulin sensitivity | Baseline to week 12
  For the calculation of this parameter the Matsuda index will be used, from the values obtained and applying the formula.
Total Cholesterol | Baseline to week 12
  The determination of total cholesterol will be made from a blood sample with the patient fasting between 8 to 12 hours. Samples will be analyzed by spectrophotometry. The result will be reported in milligrams per deciliter (mg / dL).
High-density lipoprotein (HDL) | Baseline to week 12
  The determination of HDL will be made from a blood sample with the patient fasting between 8 to 12 hours. Samples will be analyzed by spectrophotometry. The result will be reported in milligrams per deciliter (mg / dL).
Low-density lipoprotein | Baseline to week 12
  LDL will be calculated using the Friedewald formula from the results obtained of total cholesterol, HDL and triglycerides. The result will be expressed in milligrams per deciliter (mg / dl).
Triglycerides | Baseline to week 12
  The determination of triglycerides will be made from a blood sample with the patient fasting between 8 to 12 hours. Samples will be analyzed by spectrophotometry. The result will be reported in milligrams per deciliter (mg / dL).
Serum Lactate | Baseline to week 12
  The determination of serum lactate will be made from a blood sample with the patient fasting between 8 to 12 hours. Samples will be analyzed by spectrophotometry. The result will be reported in millimoles per Liter (mg / dL).

OTHER OUTCOMES:
Sleep quality | Baseline to week 12
  It will be determined by the Pittsburgh Sleep Quality Index (PSQI). This will be done by interviewing the patient and each of the components is scored. The result will be expressed in points, and a total score equal to or less than 5 will be taken as reference to determine a good sleep quality.
Tolerability to treatment | Baseline to week 12
  The patient will be instructed to record in a follow-up diary any condition, alteration or change in the state of health that could occur during the period of the intervention. In addition to this, there is the contact section where you can communicate with the investigating doctor, or protocol director to report alterations. The report of adverse effects presented as a result of the intervention will be made.
Treatment attachment | Baseline to week 12
  The attachment to treatment will be determined by quantifying remaining capsules in the bottle during monthly follow-up appointments. At the end of the study, the sum of all the capsules per medicine will be made and it will be classified as an adequate attachment to those that meet ≥ 80% of the doses during the 90 days of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lizet Yadira Rosales-Rivera, PhD Science, Principal Investigator — Instituto de terapeutica experimental y clínica
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S13-S27. doi: 10.2337/dc18-S002. PMID 29222373
- [Background] Brannick B, Wynn A, Dagogo-Jack S. Prediabetes as a toxic environment for the initiation of microvascular and macrovascular complications. Exp Biol Med (Maywood). 2016 Jun;241(12):1323-31. doi: 10.1177/1535370216654227. PMID 27302176
- [Background] Ferrannini E, Gastaldelli A, Iozzo P. Pathophysiology of prediabetes. Med Clin North Am. 2011 Mar;95(2):327-39, vii-viii. doi: 10.1016/j.mcna.2010.11.005. PMID 21281836
- [Background] Wilson ML. Prediabetes: Beyond the Borderline. Nurs Clin North Am. 2017 Dec;52(4):665-677. doi: 10.1016/j.cnur.2017.07.011. Epub 2017 Oct 5. PMID 29080583
- [Background] Hostalek U, Gwilt M, Hildemann S. Therapeutic Use of Metformin in Prediabetes and Diabetes Prevention. Drugs. 2015 Jul;75(10):1071-94. doi: 10.1007/s40265-015-0416-8. PMID 26059289
- [Background] Serrano R, Garcia-Soidan FJ, Diaz-Redondo A, Artola S, Franch J, Diez J, Carrillo L, Ezkurra P, Millaruelo JM, Segui M, Sangros FJ, Martinez-Candela J, Munoz P, Goday A, Regidor E; Grupo de Estudio PREDADS. Cohort Study in Primary Health Care on the Evolution of Patients with Prediabetes (PREDAPS): basis and methodology. Rev Esp Salud Publica. 2013 Mar-Apr;87(2):121-35. doi: 10.4321/S1135-57272013000200003. English, Spanish. PMID 23775102
- [Background] Yang H, Jin X, Kei Lam CW, Yan SK. Oxidative stress and diabetes mellitus. Clin Chem Lab Med. 2011 Nov;49(11):1773-82. doi: 10.1515/CCLM.2011.250. Epub 2011 Aug 3. PMID 21810068
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Tang WH, Martin KA, Hwa J. Aldose reductase, oxidative stress, and diabetic mellitus. Front Pharmacol. 2012 May 9;3:87. doi: 10.3389/fphar.2012.00087. eCollection 2012. PMID 22582044
- [Background] Rolo AP, Palmeira CM. Diabetes and mitochondrial function: role of hyperglycemia and oxidative stress. Toxicol Appl Pharmacol. 2006 Apr 15;212(2):167-78. doi: 10.1016/j.taap.2006.01.003. Epub 2006 Feb 20. PMID 16490224
- [Background] Brownlee M. Biochemistry and molecular cell biology of diabetic complications. Nature. 2001 Dec 13;414(6865):813-20. doi: 10.1038/414813a. PMID 11742414
- [Background] Torres-Bugarin O, Zavala-Cerna MG, Nava A, Flores-Garcia A, Ramos-Ibarra ML. Potential uses, limitations, and basic procedures of micronuclei and nuclear abnormalities in buccal cells. Dis Markers. 2014;2014:956835. doi: 10.1155/2014/956835. Epub 2014 Feb 4. PMID 24778463
- [Background] Jdey W, Thierry S, Popova T, Stern MH, Dutreix M. Micronuclei Frequency in Tumors Is a Predictive Biomarker for Genetic Instability and Sensitivity to the DNA Repair Inhibitor AsiDNA. Cancer Res. 2017 Aug 15;77(16):4207-4216. doi: 10.1158/0008-5472.CAN-16-2693. Epub 2017 Jun 6. PMID 28588010
- [Background] Kisurina-Evgenieva OP, Sutiagina OI, Onishchenko GE. Biogenesis of Micronuclei. Biochemistry (Mosc). 2016 May;81(5):453-64. doi: 10.1134/S0006297916050035. PMID 27297896
- [Background] Graham GG, Punt J, Arora M, Day RO, Doogue MP, Duong JK, Furlong TJ, Greenfield JR, Greenup LC, Kirkpatrick CM, Ray JE, Timmins P, Williams KM. Clinical pharmacokinetics of metformin. Clin Pharmacokinet. 2011 Feb;50(2):81-98. doi: 10.2165/11534750-000000000-00000. PMID 21241070
- [Background] Gong L, Goswami S, Giacomini KM, Altman RB, Klein TE. Metformin pathways: pharmacokinetics and pharmacodynamics. Pharmacogenet Genomics. 2012 Nov;22(11):820-7. doi: 10.1097/FPC.0b013e3283559b22. No abstract available. PMID 22722338
- [Background] Vecchio S, Giampreti A, Petrolini VM, Lonati D, Protti A, Papa P, Rognoni C, Valli A, Rocchi L, Rolandi L, Manzo L, Locatelli CA. Metformin accumulation: lactic acidosis and high plasmatic metformin levels in a retrospective case series of 66 patients on chronic therapy. Clin Toxicol (Phila). 2014 Feb;52(2):129-35. doi: 10.3109/15563650.2013.860985. Epub 2013 Nov 28. PMID 24283301
- [Background] Lalau JD. Lactic acidosis induced by metformin: incidence, management and prevention. Drug Saf. 2010 Sep 1;33(9):727-40. doi: 10.2165/11536790-000000000-00000. PMID 20701406
- [Background] Dunn CJ, Peters DH. Metformin. A review of its pharmacological properties and therapeutic use in non-insulin-dependent diabetes mellitus. Drugs. 1995 May;49(5):721-49. doi: 10.2165/00003495-199549050-00007. PMID 7601013
- [Background] Lardone PJ, Alvarez-Sanchez SN, Guerrero JM, Carrillo-Vico A. Melatonin and glucose metabolism: clinical relevance. Curr Pharm Des. 2014;20(30):4841-53. doi: 10.2174/1381612819666131119101032. PMID 24251676
- [Background] Brzezinski A. Melatonin in humans. N Engl J Med. 1997 Jan 16;336(3):186-95. doi: 10.1056/NEJM199701163360306. No abstract available. PMID 8988899
- [Background] Al-Omary FA. Melatonin: comprehensive profile. Profiles Drug Subst Excip Relat Methodol. 2013;38:159-226. doi: 10.1016/B978-0-12-407691-4.00005-8. PMID 23668405
- [Background] Singh M, Jadhav HR. Melatonin: functions and ligands. Drug Discov Today. 2014 Sep;19(9):1410-8. doi: 10.1016/j.drudis.2014.04.014. Epub 2014 Apr 30. PMID 24792719
- [Background] Hussain SA, Khadim HM, Khalaf BH, Ismail SH, Hussein KI, Sahib AS. Effects of melatonin and zinc on glycemic control in type 2 diabetic patients poorly controlled with metformin. Saudi Med J. 2006 Oct;27(10):1483-8. PMID 17013468
- [Background] Gamboa ML, Canales-Gómez JS, Castro Sandoval T de J. Bioavailability of Long Acting Capsules of Melatonin in Mexican Healthy Volunteers. J Bioequiv Availab. 2010 Sep 30;02(05).
- [Background] Garfinkel D, Zorin M, Wainstein J, Matas Z, Laudon M, Zisapel N. Efficacy and safety of prolonged-release melatonin in insomnia patients with diabetes: a randomized, double-blind, crossover study. Diabetes Metab Syndr Obes. 2011;4:307-13. doi: 10.2147/DMSO.S23904. Epub 2011 Aug 2. PMID 21887103
- [Background] McMullan CJ, Schernhammer ES, Rimm EB, Hu FB, Forman JP. Melatonin secretion and the incidence of type 2 diabetes. JAMA. 2013 Apr 3;309(13):1388-96. doi: 10.1001/jama.2013.2710. PMID 23549584
- [Background] Thomas AP, Hoang J, Vongbunyong K, Nguyen A, Rakshit K, Matveyenko AV. Administration of Melatonin and Metformin Prevents Deleterious Effects of Circadian Disruption and Obesity in Male Rats. Endocrinology. 2016 Dec;157(12):4720-4731. doi: 10.1210/en.2016-1309. Epub 2016 Sep 21. PMID 27653034
- [Background] Reutrakul S, Sumritsopak R, Saetung S, Chanprasertyothin S, Chailurkit LO, Anothaisintawee T. Lower nocturnal urinary 6-sulfatoxymelatonin is associated with more severe insulin resistance in patients with prediabetes. Neurobiol Sleep Circadian Rhythms. 2017 Jun 28;4:10-16. doi: 10.1016/j.nbscr.2017.06.001. eCollection 2018 Jan. PMID 31236502
- [Background] Park JH, Shim HM, Na AY, Bae KC, Bae JH, Im SS, Cho HC, Song DK. Melatonin prevents pancreatic beta-cell loss due to glucotoxicity: the relationship between oxidative stress and endoplasmic reticulum stress. J Pineal Res. 2014 Mar;56(2):143-53. doi: 10.1111/jpi.12106. Epub 2013 Nov 25. PMID 24168371
- [Background] Rybka J, Kedziora-Kornatowska K, Kupczyk D, Muszalik M, Kornatowski M, Kedziora J. Antioxidant effect of immediate- versus sustained-release melatonin in type 2 diabetes mellitus and healthy controls. Drug Deliv. 2016;23(3):814-7. doi: 10.3109/10717544.2014.917343. Epub 2014 May 28. PMID 24865293
- [Background] Lo CC, Lin SH, Chang JS, Chien YW. Effects of Melatonin on Glucose Homeostasis, Antioxidant Ability, and Adipokine Secretion in ICR Mice with NA/STZ-Induced Hyperglycemia. Nutrients. 2017 Oct 29;9(11):1187. doi: 10.3390/nu9111187. PMID 29109369
- [Background] Onaran I, Guven GS, Ozdas SB, Kanigur G, Vehid S. Metformin does not prevent DNA damage in lymphocytes despite its antioxidant properties against cumene hydroperoxide-induced oxidative stress. Mutat Res. 2006 Dec 10;611(1-2):1-8. doi: 10.1016/j.mrgentox.2006.06.036. Epub 2006 Sep 26. PMID 17000131
- [Background] Skrha J, Prazny M, Hilgertova J, Kvasnicka J, Kalousova M, Zima T. Oxidative stress and endothelium influenced by metformin in type 2 diabetes mellitus. Eur J Clin Pharmacol. 2007 Dec;63(12):1107-14. doi: 10.1007/s00228-007-0378-1. Epub 2007 Sep 15. PMID 17874238
- [Background] AIDS networking in Canada, US. CMAJ. 1995 Dec 15;153(12):1772. No abstract available. PMID 8529190